CLINICAL TRIAL: NCT07268963
Title: Biofeedback for Dysfunctional Voiding and Giggle Incontinence in Children
Brief Title: Biofeedback for Dysfunctional Voiding and Giggle Incontinence
Status: Active, not recruiting | Type: Observational
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Furkan Adem Canbaz, Medical doctor, Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital
Other Study IDs: BF DV + Giggle
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Biofeedback Therapy; Dysfunctional Voiding; Giggle Incontinence
Keywords: Giggle; Dysfunctional voiding; Incontinence; Biofeedback
MeSH Terms: interventions — Biofeedback, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Giggle incontinence: Patients who received biofeedback therapy for giggle incontinence
  Interventions: Behavioral: Biofeedback therapy
- Dysfunctional voiding: Patients who received biofeedback therapy for dysfunctional voiding
  Interventions: Behavioral: Biofeedback therapy

INTERVENTIONS:
Behavioral: Biofeedback therapy — Biofeedback therapy is a behavioral treatment method that helps patients become more aware of and gain better control over their pelvic floor muscles. Using EMG electrodes, muscle activity is monitored and presented to the patient visually or audibly, enabling them to recognize and correct improper muscle contractions or relaxations that contribute to urinary incontinence.

SUMMARY:
This study aims to evaluate the efficacy of biofeedback treatment for dysfunctional voiding and giggle incontinence in children. Predictive factors of treatment success will also researched.

DETAILED DESCRIPTION:
A total of approximately 60 patients who received biofeedback therapy will be evaluated retrospectively. Treatment success rates among these patients will be evaluated. Patients will be divided into mainly two groups according to the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with dysfunctional voiding or giggle incontinence
* Patients treated with biofeedback therapy

Exclusion Criteria:

* Presence of anatomical or neurological problems
* Patients with missing data

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who were received biofeedback therapy for dysfunctional voiding and giggle incontinece in pediatric urology clinic of Sancaktepe Sehit Prof Dr Ilhan Varank Training and Research Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Biofeedback-Related Resolution | From enrollment to the end of treatment at 18 weeks
  Participants achieved a complete response which means 100% improvement in resolution of incontinence and abnormal voiding pattern

OTHER OUTCOMES:
Predictive Factors of Treatment Response | 18 weeks
  Age, gender, and diagnosis will be evaluated as potential predictive factors of treatment response

CONTACTS AND LOCATIONS:
Locations (1):
- Sancaktepe Sehit Prof dr Ilhan Varank Training and Research Hospital, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I do not have any idea.

REFERENCES:
- [Background] Sadeghi M, Oskouie IM, Naserghandi A, Arvin A, Majidi Zolbin M. Exploring dysfunctional voiding in girls: a comprehensive literature review of assessment and management strategies. BMC Urol. 2025 Apr 12;25(1):87. doi: 10.1186/s12894-025-01772-0. PMID 40221717
- [Background] Gonzalez-Maldonado AA, Garcia-Merida M. Giggle incontinence: a scoping review. Pediatr Res. 2024 Jun;95(7):1720-1725. doi: 10.1038/s41390-024-03065-y. Epub 2024 Feb 2. PMID 38307925